CLINICAL TRIAL: NCT03478267
Title: The Relationship Between Fetal Baseline Heart-rate and the Level of Acetyl-choline Esterase in Fetal Blood
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Vered Lamhot MD, Primary investigator, Rambam Health Care Campus
Other Study IDs: 0584-16-RMB
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Fetal Heart Failure (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal heart rate 110-130 bpm: Pregnancies in which the fetal baseline heart rate is between 110 beats per minute and 130 beats per minute.
  Interventions: Diagnostic Test: AChE levels
- Fetal heart rate 140-160 bpm: Pregnancies in which the fetal baseline heart rate is between 140 beats per minute and 160 beats per minute.
  Interventions: Diagnostic Test: AChE levels

INTERVENTIONS:
Diagnostic Test: AChE levels — AChE levels in peripheral blood tests from maternal blood, fetal umbilical cord and placenta.

SUMMARY:
Pregnant women between 32-41 weeks' gestation designated for either vaginal birth or cesarean section will be recruited for the study. Data regarding maternal resting heart rate and fetal baseline heart rate as depicted on the monitor will be collected. A blood sample will be acquired from the parturient and the umbilical cord as well as a sample from the placenta will be obtained. Levels of Acetyl Choline Esterase (AChE) will be determined from all aforementioned samples. Statistical correlation between fetal baseline heart rate and fetal and maternal AChE levels will be assessed.

DETAILED DESCRIPTION:
Pregnant women between 32-41 weeks' gestation designated for either vaginal birth or cesarean section will be recruited for the study. After signing an informed consent, data regarding maternal resting heart rate and fetal baseline heart rate as depicted on the monitor will be collected.

Patients will be divided into 2 equal groups according to fetal baseline heart rate:

1. st group-fetal heart rate between 110-130 beats per minute (bpm).
2. nd group-fetal heart rate between 140-160 bpm. A blood sample will be acquired from the parturient and the umbilical cord as well as a sample from the placenta will be obtained. Levels of Acetyl Choline Esterase (AChE) will be determined from all aforementioned samples. Statistical correlation between fetal baseline heart rate and fetal and maternal AChE levels will be assessed.

Data regarding demographic, medical and obstetric information of the participants will be obtained from the hospital's electronic records.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 32 and 41 weeks' gestation undergoing either vaginal or cesarean delivery with a fetal baseline heart rate of 110-130 beats per minute and 140-160 beats per minute.

Exclusion Criteria:

1. Delivery before 32 weeks of gestation
2. Maternal bradycardic (<60) or tachycardic (>100) resting heart rate.
3. Fetal bradycardia (<110) or tachycardia (>160).
4. Suspected chorioamnionitis
5. Maternal diseases which can affect her heart rate such as:

   1. Cardiac disease (including arrhythmias)
   2. Diseases of the thyroid gland
   3. Rheumatic diseases
6. Use of medication which alters heart rate such as:

   1. Beta blockers
   2. Beta agonists
   3. Cocaine, amphetamines
7. Use of Pethidine and Phenergan during delivery

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female pregnant patients and their fetuses
Study Population: Pregnant women between 32 and 41 weeks' gestation undergoing either vaginal or cesarean delivery with a fetal baseline heart rate of 110-130 beats per minute and 140-160 beats per minute.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-02-17 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
AChE levels in fetal blood | Up to 5 minutes post delivery (either vaginal or cesarean)
  AChE levels obtained from the fetal umbilical cord after birth

SECONDARY OUTCOMES:
AChE levels in maternal blood | Up to 5 minutes post delivery (either vaginal or cesarean)
  AChE levels obtained from maternal peripheral blood after birth
AChE levels in the placenta | Up to 30 minutes post delivery (either vaginal or cesarean)
  AChE levels obtained from the placenta after birth

CONTACTS AND LOCATIONS:
Overall Officials: Vered Lamhot, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam hospital, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided